CLINICAL TRIAL: NCT04695847
Title: A Phase I Open Label First in Human Dose Escalation and Expansion Study of the Bispecific Anti-Mucin 1 - Epidermal Growth Factor Receptor Antibody Drug Conjugate M1231 as a Single Agent in Participants With Advanced Solid Tumors
Brief Title: M1231 in Participants With Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: EMD Serono Research & Development Institute, Inc. (Industry)
Collaborators: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Organization: EMD Serono (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MS201668_0001
Record Dates: First submitted 2021-01-04; First posted 2021-01-05 (Actual); Last update posted 2023-07-07 (Actual); Status verified 2023-07

CONDITIONS: Metastatic Solid Tumors; Esophageal Cancer; Non-Small Cell Lung Cancer
Keywords: M1231; Non-Small Cell Lung Cancer; Metastatic Solid Tumors; Esophageal cancer; Maximum tolerated dose; Pharmacokinetics
MeSH Terms: conditions — Esophageal Neoplasms; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part 1: M1231 (Experimental): Participants with solid tumors for whom no effective standard therapy exists will be included in this Part. Dose escalation of M1231 will be administered as single agent.
  Interventions: Drug: M1231
- Part 2: Cohort A M1231: Metastatic NSCLC (Experimental): Participants with metastatic Non-small Cell Lung Cancer (NSCLC) expressing Epidermal Growth Factor Receptor (EGFR) and Mucin 1 (MUC1) on archival tumor tissue will receive M1231 at the dose determined as recommended dose for expansion (RDE) in Part 1.
  Interventions: Drug: M1231
- Part 2: Cohort B M1231: Metastatic Esophageal Squamous Cell Carcinoma (Experimental): Participants with metastatic esophageal squamous cell carcinoma will receive M1231 at the dose determined as recommended dose for expansion (RDE) in Part 1.
  Interventions: Drug: M1231

INTERVENTIONS:
Drug: M1231 — M1231 will be administered at escalated doses every three weeks until disease progression, unacceptable toxicity, withdrawal of consent, or any criterion for withdrawal from the study.
  Other Names: Bispecific antibody drug conjugate (ADC)
  Arms: Part 1: M1231
Drug: M1231 — M1231 will be administered at the dose determined as RDE in part 1, every three weeks until disease progression, unacceptable toxicity, withdrawal of consent, or any criterion for withdrawal from the study.
  Other Names: Bispecific antibody drug conjugate (ADC)
  Arms: Part 2: Cohort A M1231: Metastatic NSCLC; Part 2: Cohort B M1231: Metastatic Esophageal Squamous Cell Carcinoma

SUMMARY:
This study is to establish a safe and tolerable dose and to investigate pharmacokinetics and the first clinical efficacy signals of M1231 as a single agent in participants with solid tumors (Part 1) and with metastatic Non-small Cell Lung Cancer (NSCLC) and esophageal squamous cell carcinoma (Part 2). Dose escalation will be followed by the dose expansion once the maximum tolerated dose (MTD) or recommended dose for Expansion (RDE) has been defined.

ELIGIBILITY:
Inclusion Criteria:

For Part 1 and 2:

* The Investigator reviews the medical history, menstrual history, and recent sexual activity to decrease the risk for inclusion of a female with an early undetected pregnancy

For Part 1:

* Locally advanced or metastatic disease that is intolerant or refractory to standard therapy or for which no standard therapy is judged appropriate by the investigator
* Participants with solid tumors expressing or likely to expressing EGFR and MUC1, including but not limited to lung cancer, squamous esophageal cancer, head and neck squamous cell carcinoma, breast cancer and ovarian cancer, should be prioritized for enrollment

For Part 2:

* Cohort A: Participants must have progressed on at least 2 prior lines of therapy
* Cohort B: Participants must have progressed on at least 1 prior line of platinum therapy and for microsatellite instability-high (MSI-H) at least 1 prior line with pembrolizumab
* Eastern Cooperative Oncology Group (ECOG) Performance Status less than 1
* Tumor accessible for biopsies and agreement to conduct fresh tumor biopsies at Screening and before first dosing

Exclusion Criteria:

* Participants not recovered from adverse events (AE) (less than or equal to Grade 1) related to previous therapies (excluding Grade 1 neuropathy and alopecia)
* Participant has a history of a second malignancy within 3 years before the date of enrollment
* Known brain metastasis
* Unstable angina, myocardial infarction, congestive heart failure or a coronary revascularization procedure within 180 days of study entry
* Cerebrovascular accident/stroke
* Diagnosis of fever within 1 week prior to study intervention administration
* Life expectancy of less than 4 months
* Steroid therapy for anti-neoplastic intent taken less than 7 days prior to the first dose of study intervention
* Major surgery within 4 weeks prior to start of study intervention
* Received growth factors (including erythropoietin (EPO), darbepoetin, granulocyte-colony stimulating factor (G-CSF), granulocyte macrophage-colony stimulating factor (GM-CSF), and platelet stimulators or transfusions within 2 weeks prior to the first day of study intervention

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2021-01-13 (Actual); Primary Completion 2023-06-23 (Actual); Study Completion 2023-06-23 (Actual)

PRIMARY OUTCOMES:
Part 1: Number of Participants with Dose Limiting Toxicities (DLTs) | Day 1 Up to Day 21
Part 1: Number of Participants with Treatment Emergent Adverse Events (TEAEs) and Treatment Related TEAEs | From Baseline until 4 months
Part 2: Objective Response (OR) According to Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1 as Assessed by Investigators | From Baseline until 6 months
Part 2: Number of Participants with Treatment Emergent Adverse Events (TEAEs) and Treatment Related TEAEs | From Baseline until 6 months
Part 2: Duration of Response (DoR) According to Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1 as Assessed by Investigators | From Baseline until 6 months

SECONDARY OUTCOMES:
Part 1:Area Under Plasma Concentration-Time Curve Within One Dosing Interval (AUC0-tau) of M1231 (Conjugated Payload), Total Antibody and Free Payload M1231 | Cycle 1 Day 1 to Cycle 3 Day 15 and every second cycle from Cycle 4 (each cycle is of 21 days), assessed up to approximately 4 months
Part 1: Dose Normalized Area Under Concentration-Time Curve Within One Dosing Interval (AUC0-tau/Dose) of M1231 (Conjugated Payload), Total Antibody and Free Payload for M1231 | Cycle 1 Day 1 to Cycle 3 Day 15 and every second cycle from Cycle 4 (each cycle is of 21 days), assessed up to approximately 4 months
Part 1: Area Under the Concentration-time Curve From Time Zero to the Last Sampling time (AUC 0-tlast) of M1231 (Conjugated Payload), Total Antibody and Free Payload for M1231 | Cycle 1 Day 1 to Cycle 3 Day 15 and every second cycle from Cycle 4 (each cycle is of 21 days), assessed up to approximately 4 months
Part 1: Dose Normalized Area Under Concentration-Time Curve From Time Zero to the Last Sampling Time (AUC0-last/Dose) of M1231 (Conjugated Payload), Total Antibody and Free Payload | Cycle 1 Day 1 to Cycle 3 Day 15 and every second cycle from Cycle 4 (each cycle is of 21 days), assessed up to approximately 4 months
Part 1: Area Under the Plasma Concentration-Time Curve From Time Zero to Infinity (AUC0-inf) of M1231 (Conjugated Payload), Total Antibody and Free Payload for M1231 | Cycle 1 Day 1 to Cycle 3 Day 15 and every second cycle from Cycle 4 (each cycle is of 21 days), assessed up to approximately 4 months
Part 1: Dose Normalized Area Under Concentration-Time Curve From Time Zero (dosing time) Extrapolated to Infinity (AUC0-inf/Dose) of M1231 (Conjugated Payload), Total Antibody and Free Payload for M1231 | Cycle 1 Day 1 to Cycle 3 Day 15 and every second cycle from Cycle 4 (each cycle is of 21 days), assessed up to approximately 4 months
Part 1: Area Under Concentration From Time tlast Extrapolated to Infinity (AUCextra%) of M1231 (Conjugated Payload), Total Antibody and Free Payload for M1231 | Cycle 1 Day 1 to Cycle 3 Day 15 and every second cycle from Cycle 4 (each cycle is of 21 days), assessed up to approximately 4 months
Part 1: Observed Concentration At The End of The Infusion Period (Ceoi) of M1231 (Conjugated Payload), Total Antibody and Free Payload for M1231 | Cycle 1 Day 1 to Cycle 3 Day 15 and every second cycle from Cycle 4 (each cycle is of 21 days), assessed up to approximately 4 months
Part 1: Total Body Clearance (CL) of M1231 (Conjugated Payload), Total Antibody and Free Payload for M1231 | Cycle 1 Day 1 to Cycle 3 Day 15 and every second cycle from Cycle 4 (each cycle is of 21 days), assessed up to approximately 4 months
Part 1: Plasma Concentration Observed Immediately Before Next Dosing (Ctrough) of M1231 (Conjugated Payload), Total Antibody and Free Payload for M1231 | Cycle 1 Day 1 to Cycle 3 Day 15 and every second cycle from Cycle 4 (each cycle is of 21 days), assessed up to approximately 4 months
Part 1: Accumulation Ratio for AUCtau (Racc[AUCtau]) of M1231 (Conjugated Payload), Total Antibody and Free Payload for M1231 | Cycle 1 Day 1 to Cycle 3 Day 15 and every second cycle from Cycle 4 (each cycle is of 21 days), assessed up to approximately 4 months
Part 1: Accumulation Ratio for Maximum Observed Concentration (Racc[Cmax]) of M1231 (Conjugated Payload), Total Antibody and Free Payload for M1231 | Cycle 1 Day 1 to Cycle 3 Day 15 and every second cycle from Cycle 4 (each cycle is of 21 days), assessed up to approximately 4 months
Part 1: Apparent Terminal Half-life (t1/2) of M1231 (Conjugated Payload), Total Antibody and Free Payload for M1231 | Cycle 1 Day 1 to Cycle 3 Day 15 and every second cycle from Cycle 4 (each cycle is of 21 days), assessed up to approximately 4 months
Part 1: Time to Reach Maximum Plasma Concentration (tmax) of M1231 (Conjugated Payload), Total Antibody and Free Payload for M1231 | Cycle 1 Day 1 to Cycle 3 Day 15 and every second cycle from Cycle 4 (each cycle is of 21 days), assessed up to approximately 4 months
Part 1: Apparent Volume of Distribution During Terminal Phase Following Extravascular Administration (Vz) of M1231 (Conjugated Payload), Total Antibody and Free Payload for M1231 | Cycle 1 Day 1 to Cycle 3 Day 15 and every second cycle from Cycle 4 (each cycle is of 21 days), assessed up to approximately 4 months
Part 1: Number of Participants with Corrected QT Interval (QTc) | Cycle 1 Day 1 to Cycle 3 Day 8 (each Cycle is of 21 days)
Part 1: Number of Participants With Anti-Drug Antibodies (ADA) against M1231 | From Baseline until 4 months
Part 1: Levels of Titers of Anti-Drug Antibody (ADA) against M1231 | From Baseline until 4 months
Part 1: Level of Mucin 1 (MUC1) Protein Expression in Archival Tumor Tissue Determined by Assay | From Baseline until 4 months
Part 1: Level of Epidermal Growth Factor Receptor (EGFR) Protein Expression in Archival Tumor Tissue Determined by Assay | From Baseline until 4 months
Part 1: Renal Clearance of Unconjugated Hemiasterlin Analogue (a tubulin inhibitor in tumor cells) | From Baseline until 4 months
Part 1:Objective Response (OR) According to Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1 as Assessed by Investigators | From Baseline until 4 months
Part 1: Duration of Response (DoR) According to Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1 as Assessed by Investigators | From Baseline until 4 months
Part 1: Progression-free survival (PFS) According to Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1 as Assessed by Investigators | From Baseline until 4 months
Part 2: Progression-free survival (PFS) According to Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1 as Assessed by Investigators | From Baseline until 6 months
Part 2: Overall Survival (OS) According to Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1 as Assessed by Investigators | From Baseline until 6 months
Part 2: Level of Mucin 1 (MUC1) Protein Expression in Archival Tumor Tissue Determined by Assay | From Baseline until 6 months
Part 2: Level of Epidermal Growth Factor Receptor (EGFR) Protein Expression in Archival Tumor Tissue Determined by Assay | From Baseline until 6 months
Part 2: Area Under Plasma Concentration-Time Curve Within One Dosing Interval (AUC0-tau) of M1231 (Conjugated Payload), Total Antibody and Free Payload M1231 | Cycle 1 Day 1 to Cycle 3 Day 3 and every second cycle from Cycle 4 (each cycle is of 21 days), assessed up to approximately 6 months
Part 2: Dose Normalized Area Under Concentration-Time Curve Within One Dosing Interval (AUC0-tau/Dose) of M1231 (Conjugated Payload), Total Antibody and Free Payload for M1231 | Cycle 1 Day 1 to Cycle 3 Day 3 and every second cycle from Cycle 4 (each cycle is of 21 days), assessed up to approximately 6 months
Part 2:Area Under the Concentration-time Curve From Time Zero to the Last Sampling time (AUC 0-tlast) of M1231 (Conjugated Payload), Total Antibody and Free Payload for M1231 | Cycle 1 Day 1 to Cycle 3 Day 3 and every second cycle from Cycle 4 (each cycle is of 21 days), assessed up to approximately 6 months
Part 2: Dose Normalized Area Under Concentration-Time Curve From Time Zero to the Last Sampling Time (AUC0-last/Dose) of M1231 (Conjugated Payload), Total Antibody and Free Payload for M1231 | Cycle 1 Day 1 to Cycle 3 Day 3 and every second cycle from Cycle 4 (each cycle is of 21 days), assessed up to approximately 6 months
Part 2:Area Under the Plasma Concentration-Time Curve From Time Zero to Infinity (AUC0-inf) of M1231 (Conjugated Payload), Total Antibody and Free Payload for M1231 | Cycle 1 Day 1 to Cycle 3 Day 3 and every second cycle from Cycle 4 (each cycle is of 21 days), assessed up to approximately 6 months
Part 2:Dose Normalized Area Under Concentration-Time Curve From Time Zero (dosing time) Extrapolated to Infinity (AUC0-inf/Dose) of M1231 (Conjugated Payload), Total Antibody and Free Payload for M1231 | Cycle 1 Day 1 to Cycle 3 Day 3 and every second cycle from Cycle 4 (each cycle is of 21 days), assessed up to approximately 6 months
Part 2:Area Under Concentration From Time tlast Extrapolated to Infinity (AUCextra%) of M1231 (Conjugated Payload), Total Antibody and Free Payload for M1231 | Cycle 1 Day 1 to Cycle 3 Day 3 and every second cycle from Cycle 4 (each cycle is of 21 days), assessed up to approximately 6 months
Part 2:Observed Concentration At The End of The Infusion Period (Ceoi) of M1231 (Conjugated Payload), Total Antibody and Free Payload for M1231 | Cycle 1 Day 1 to Cycle 3 Day 3 and every second cycle from Cycle 4 (each cycle is of 21 days), assessed up to approximately 6 months
Part 2: Total Body Clearance (CL) of M1231 (Conjugated Payload), Total Antibody and Free Payload for M1231 | Cycle 1 Day 1 to Cycle 3 Day 3 and every second cycle from Cycle 4 (each cycle is of 21 days), assessed up to approximately 6 months
Part 2:Plasma Concentration Observed Immediately Before Next Dosing (Ctrough) of M1231 (Conjugated Payload), Total Antibody and Free Payload for M1231 | Cycle 1 Day 1 to Cycle 3 Day 3 and every second cycle from Cycle 4 (each cycle is of 21 days), assessed up to approximately 6 months
Part 2:Accumulation Ratio for AUCtau (Racc[AUCtau]) of M1231 (Conjugated Payload), Total Antibody and Free Payload for M1231 | Cycle 1 Day 1 to Cycle 3 Day 3 and every second cycle from Cycle 4 (each cycle is of 21 days), assessed up to approximately 6 months
Part 2:Accumulation Ratio for Maximum Observed Concentration (Racc[Cmax]) of M1231 (Conjugated Payload), Total Antibody and Free Payload for M1231 | Cycle 1 Day 1 to Cycle 3 Day 3 and every second cycle from Cycle 4 (each cycle is of 21 days), assessed up to approximately 6 months
Part 2:Apparent Terminal Half-life (t1/2) of M1231 (Conjugated Payload), Total Antibody and Free Payload for M1231 | Cycle 1 Day 1 to Cycle 3 Day 3 and every second cycle from Cycle 4 (each cycle is of 21 days), assessed up to approximately 6 months
Part 2:Time to Reach Maximum Plasma Concentration (tmax) of M1231 (Conjugated Payload), Total Antibody and Free Payload for M1231 | Cycle 1 Day 1 to Cycle 3 Day 3 and every second cycle from Cycle 4 (each cycle is of 21 days), assessed up to approximately 6 months
Part 2:Apparent Volume of Distribution During Terminal Phase Following Extravascular Administration (Vz) of M1231 (Conjugated Payload), Total Antibody and Free Payload for M1231 | Cycle 1 Day 1 to Cycle 3 Day 3 and every second cycle from Cycle 4 (each cycle is of 21 days), assessed up to approximately 6 months
Part 2:Number of Participants with Anti-Drug Antibodies (ADA) against M1231 | From Baseline until 6 months
Part 2: Levels of Titers of Anti-Drug Antibody (ADA) against M1231 | From Baseline until 6 months
Part 2: Number of Participants with Corrected QT Interval (QTc) | Cycle 1 Day 1 to Cycle 3 Day 8 (each Cycle is of 21 days)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck Healthcare KGaA, Darmstadt, Germany, an affiliate of Merck KGaA, Darmstadt, Germany
Locations (3):
- United States (2):
  - MD Anderson Cancer Center - Clinical Cancer Prevention, Houston, Texas
  - NEXT Oncology, San Antonio, Texas
- Princess Margaret Cancer Centre, Toronto, Canada

IPD SHARING:
Plan to Share IPD: No
We are committed to enhancing public health through responsible sharing of clinical trial data. Following approval of a new product or a new indication for an approved product in both the US and the European Union, the study sponsor and/or its affiliated companies will share study protocols, anonymized patient data and study level data, and redacted clinical study reports with qualified scientific and medical researchers, upon request, as necessary for conducting legitimate research. Further information on how to request data can be found on our website https://bit.ly/IPD21

REFERENCES:
- See also: Trial Awareness and Transparency website — https://clinicaltrials.emdgroup.com/en/trial-details/?id=MS201668_0001
- See also: US Medical Information website, Medical Resources — https://medical.emdserono.com/en_US/home.html